CLINICAL TRIAL: NCT05216068
Title: Investigation and Diagnosis of the Chromosome Variation in Donated/abandoned Blastocyst
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CMRPG8M0241
Record Dates: First submitted 2022-01-23; First posted 2022-01-31 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Chromosome Translocation; Genetic Disorders in Pregnancy; Recurrent Miscarriage
Keywords: pre-implantation genetic diagnosis; balanced reciprocal translocation (BRT); structural variation (SV); next generation sequencing; abandoned blastocysts
MeSH Terms: conditions — Translocation, Genetic; Abortion, Habitual

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- donated abandonment embryos (Other): Embryos biopsies for PGT-A (by use of NGS platforms from our institute) will be used for the validation of our Lab QC.
  Interventions: Diagnostic Test: NGS

INTERVENTIONS:
Diagnostic Test: NGS — Based on the next generation sequencing (NGS), WES can identify single nucleotide variants (SNVs) and small variants.

SUMMARY:
Blastocysts derived from patients seeking infertility treatment were generated by in vitro fertilization and embryo culture as previously described, and were evaluated using the Gardner system. As part of the embryo selection process, cells of TE biopsy were collected, and blastocysts were vitrified. The clinical TE biopsies were subjected to whole genome amplification (WGA) with SurePlex reagents (Illumina) followed by NGS-based PGT-A using Illumina's VeriSeq kit (Illumina) on a MiSeq system (Illumina) according to the manufacturer's protocol.

DETAILED DESCRIPTION:
Collected 200 donate abandonment embryos (well-developed blastocysts) for research under the National Assisted Reproduction Act of Taiwan.

1. Collected 200 donate abandonment embryos: Five to six days after egg retrieval, well-developed embryos (called blastocysts).
2. Blastocysts derived from patients seeking infertility treatment were generated.
3. Embryos biopsies for PGT-A (by use of NGS platforms from our institute) will be used for the validation of our Lab QC embryo.
4. To standardize the operating procedures
5. Paper writing.

ELIGIBILITY:
Inclusion Criteria:

* the surplus blastocysts
* parents consent to donate the embryos

Exclusion Criteria:

* not agree to participate in this program
* whose embryo morphology and quality do not meet the technical requirements for genetic testing

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Blastocyst aneuploidy rate | 28 days
  anormal Karyotype according to human genome 19 or updated version

SECONDARY OUTCOMES:
Whole genome amplification rate | 7 days
  success rate

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan